CLINICAL TRIAL: NCT06460116
Title: Health Equity and Rural Education (HERE!) Clinical Trial: A Healthcare-Community Partnership Leveraging School-Based Community Health Workers to Improve Student Attendance
Brief Title: Health Equity and Rural Education (HERE!) Clinical Trial
Acronym: HERE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00151155; 1R56NR021161-01 (NIH)
Record Dates: First submitted 2024-02-06; First posted 2024-06-14 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Behavioral Symptoms; Community Health Workers; Social Determinants of Health; Educational Problems
MeSH Terms: conditions — Behavioral Symptoms | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This is a two phase feasibility pilot. Consistent with the community engaged approach, the first study phase is interviews with at least 30 stakeholders to enhance the school-based community health worker (SB-CHW) intervention and the enhanced usual care (EUC) arms. The second study phase is a feasibility trial to assess the feasibility of the SB-CHW condition across 38 students and 38 parent/guardians and the EUC condition across 10 students and their 10 parents/guardians.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study Phase I: Stakeholder Interviews (No Intervention): Phase I interviews with stakeholders (Community Advisory Board members, CHWs, community members, students Grade 6-12, & parent stakeholders) will be completed to inform the school-based community health worker and the enhanced usual care conditions in the Phase 2 feasibility pilot.
- Study Phase II: School-based Community Health Worker Intervention (Experimental): The School-Based Community Health Worker (SB-CHW) intervention is the active intervention in the Phase II feasibility trial.
  Interventions: Behavioral: School-Based Community Health Worker (SB-CHW) intervention
- Study Phase II: Enhanced Usual Care (Active Comparator): Enhanced usual care (EUC) is the comparator in the Phase II feasibility trial.
  Interventions: Behavioral: Enhanced Usual Care (EUC) Methods

INTERVENTIONS:
Behavioral: School-Based Community Health Worker (SB-CHW) intervention — The school-based community health worker will support students with chronic poor attendance and their parent/guardian for a minimum of two 30-minute encounters focused on addressing social determinants needs, understanding the range/student encounter varies greatly due to the intensity of the social need(s) (e.g., crisis/noncrisis) and the number of needs being jointly addressed. The SB-CHW will build relationships across encounters and apply trauma-informed best practices.
  Arms: Study Phase II: School-based Community Health Worker Intervention
Behavioral: Enhanced Usual Care (EUC) Methods — The network of school-based health centers without school-based community health workers will receive reminders of the the existing online social services directory.
  Arms: Study Phase II: Enhanced Usual Care

SUMMARY:
The goal of this community-engaged research is two-fold. The first goal is to gather stakeholder feedback to inform a school-based community health worker intervention with youth with poor school attendance and an enhanced usual care condition. The second goal is to evaluate the feasibility of implementing the school-based community health worker intervention and enhanced usual care approach within rural schools.

The main question it aims to answer is whether it is feasibile to recruit children with poor school attendance and their families to the intervention, to complete the trauma-informed intervention, and to complete the associated study measures of meeting social determinants of health/mental health needs, school-based health center utilization, and behavioral helath symptoms. At least 38 rural students in grades 6-12 with poor school attendance and their parents/guardians will meet with the school-based community health worker for support around social determinants of health needs that may be barriers to attendance. Researchers will also assess the feasibility of recruiting at least 10 rural students and their parents/guardians to complete the study measures in an enhanced usual care condition in which the school-based health center without a school-based community health worker is reminded of the availability of an online social services directory.

DETAILED DESCRIPTION:
The HERE pilot study will consist of two phases to strengthen and finalize the HERE school-based community health worker (SB-CHW) intervention. The 6-month Phase I will provide broad stakeholder feedback on the proposed model and rationale, the SB-CHW intervention, the associated domains and measures, and the evaluation. The following 18-month Phase II will align with the school year and provide a feasibility test of the training, intervention, data collection, and analyses.

ELIGIBILITY:
Phase I Stakeholder Interviews (nonintervention):

Inclusion Criteria:

* A member of the program's Community Advisory Board, including community health workers;
* Caregiver of a child ages 12-18 from the Southeast Kansas region; or
* Student at least 12 years in age.

Phase II Feasibility Pilot- SB-CHW Intervention and Enhanced Usual Care Conditions

Inclusion Criteria:

* Children ages 12-18 and their parents/guardians from the Southeast Kansas region
* Student with or at risk for chronic poor attendance (missing 10% or more of the days that school has been in session at any point in the school year)

Exclusion Criteria:

* Parents/guardians or youth with profound intellectual/cognitive disability will be excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
School Based Health Services Utilization | At study completion (an average of 10 months/1 school year)
  The number of visits to School Based Health Centers (SBHC)
School Attendance | At study completion (an average of 10 months/1 school year)
  The number of school days in attendance, collected by ½ day increments
  1(b) determination whether the student continues to meet the definition of chronic poor attendance (Yes/No)

SECONDARY OUTCOMES:
Parent & Child Self-Sufficiency and Needs | At enrollment, at study completion (an average of 10 months/1 school year)
  Arizona Self-Sufficiency Matrix. An 18-item self-report measure assessing needs on a 5-point Likert scale, including Housing, Employment, Income, Food, Childcare, Children's Education, Adult Education, Health Care Coverage, Life Skills, Family/Social Relations, Mobility, Community Involvement, Parenting Skills, Legal, Mental Health, Substance Abuse, Safety, and Disabilities.
Child and Adolescent Needs and Strengths | At enrollment, at study completion (an average of 10 months/1 school year)
  Child and Adolescent Needs and Strengths (CANS) is a validated semi-structured interview that assesses children's exposure to potentially traumatic experiences & level of traumatic stress symptoms, as well as considering strengths (Kisiel & Fehrenbach, 2015).
Family Engagement | At enrollment, at study completion (an average of 10 months/1 school year)
  The Family Engagement Survey -- Version 2 (FES), a validated measure of family and school engagement consisting of 20 items rated on a Likert-type scale from 1 (Strongly Disagree) to 5 (Strongly Agree).
School-Based Community Health Worker Interactions | At study completion (an average of 10 months/1 school year)
  Number of CHW interactions with the student, parent/guardian, and/or both
Process for Enhanced Usual Care | At enrollment, at study completion (an average of 10 months/1 school year)
  Use of resources from the online social services directory (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Eve-Lynn Nelson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the Data Sharing for Demographic Research (DSDR) data repository hosted at ICPSR. Datasets in DSDR will be findable and identifiable through a study digital object identifier (DOI) minted by ICPSR. Monitoring of and compliance with this Data Management and Sharing Plan will be the responsibility of the project's Principal Investigator and follow the data management and sharing plan compliance system through The Office of Sponsored Programs at the University of Kansas Medical Center that will be administering this award. The Office of Sponsored Programs will also look for the funder requirements and will include that information in the annual progress report.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Final submission and release of the study data will occur approximately 6 months following the end of Phase 1 and Phase 2, respectively, and within the award period. Study data deposited in DSDR will be available to the research community in perpetuity. Datasets underlying methodological publications will be shared at or prior to initial publication date.
Access Criteria: All deidentified study data that are not designated as restricted use will be made available as public use data to the research community via DSDR, with users of the public use data compliant with all Terms of Use. Data that are determined to be potentially identifying through indirect or deductive disclosure are provided under restricted data contract to users who demonstrate a valid research need and meet conditions of use. Access to restricted study data is available via a virtual data enclave system at DSDR/ICPSR.